CLINICAL TRIAL: NCT02391831
Title: Prospective Study of the Natural History of Patients With Type 2 and 3 Spinal Muscular Atrophy
Acronym: NatHis-SMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Collaborators: Institut Roche (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NatHis-SMA; IDRCB-2014-A01263-44 (Other: ANSM (French Regulatory Authority))
Record Dates: First submitted 2015-03-02; First posted 2015-03-18 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Spinal Muscular Atrophy; Type 3 Spinal Muscular Atrophy
Keywords: SMA; Spinal Muscular Atrophy; Neuromuscular disease
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal; Neuromuscular Diseases | interventions — Functional Status; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Strength, function and activity measurements
Other: Muscle MRI
Other: Electrophysiology measurements
Other: Blood sampling for biomarker analysis

SUMMARY:
NatHis-SMA is a prospective, longitudinal and interventional study of the natural history of patients with type 2 and 3 Spinal Muscular Atrophy (SMA). The purpose of this study is to characterize the disease course over 2 years and identify prognostic variables of the disease and biomarkers of SMA progression, as well as determine the best outcome measures for further therapeutics approaches.

ELIGIBILITY:
INCLUSION CRITERIA

* Type 2 or 3 spinal muscular atrophy genetically confirmed
* Age superior or equal to 2 years old up to 30 years of age included
* For patients older than 6 years old, willing and able to comply with all protocol requirements and procedures.
* For non-ambulant patients, able to sit upright in a wheelchair for at least three hours
* Patients over 18 years of age and parent(s)/legal guardian(s) of patients < 18 years of age must provide written informed consent prior to participating in the study and informed assent will be obtained from minors at least 7 years of age when required by regulation.
* In France only: Affiliated to or a beneficiary of a social security category

EXCLUSION CRITERIA

* Previously treated with an investigational drug within 6 months prior the recruitment in this study.
* Other condition which may significantly interfere with the assessment of the SMA and is clearly not related to the disease
* Current or anticipated participation in any therapeutic investigational clinical studies.
* Patients with specific contraindication to MRI (i.e. metallic foreign body, claustrophobia, and others deemed to be prohibitive by the investigators) will be allowed to participate, but MRI will not be performed.
* For women : pregnancy or current breastfeeding

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of muscle strength | Baseline and then every 6 months until end of the study, up to 24 months
  Study-specific assessments: Grip and pinch strength
Change from baseline of motor function | Baseline and then every 6 months until end of the study, up to 24 months
  Study-specific assessments: Moviplate and MFM scores, upper extremity functional reaching volume, timed tests (time to rise from floor, time to walk 10 meters, time to climb and descend stairs, distance walked on the Six-Minute Walk Test)

SECONDARY OUTCOMES:
Change from baseline of respiratory function | Baseline and then every 6 months until end of the study, up to 24 months
  Study-specific assessments: Pulmonary function tests
Change from baseline of physical activity of upper limbs movements | Baseline and then every 6 months until end of the study, up to 24 months
  Quantity and duration of movements, time of inactivity during the day
Change from baseline of skeletal muscle nuclear magnetic resonance (NMR) imaging (MRI) | Baseline and then every 12 months until the end of the study, up to 24 months
  Muscle volume changes, intramuscular fatty infiltration progression, indices of disease activity (only for Paris and Strasbourg sites and for patients older than 4 years)
Change from baseline of electrophysiology measurements | Baseline and then every 6 months until end of the study, up to 24 months
  Compound Motor Action Potential (CMAP) Amplitude and Decrement search
Change from baseline of Biomarkers of SMA progression | Baseline and then every 6 months until end of the study, up to 24 months
  SMN mRNA and protein analysis, SMA exploratory biomarkers (e.g. mRNA, DNA profiling, RNA profiling, proteomic profiling)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, Principal Investigator — Association Institut de Myologie
Locations (9):
- Belgium (2):
  - Reference centre for neuromuscular diseases - UZ Leuven - Department of Pediatrics - University Hospitals Leuven, Leuven
  - Centre de Référence neuromusculaire - CHR La Citadelle, Liège
- France (6):
  - Service de Rééducation Pédiatrique Infantile " L'Escale " - Hôpital Femme Mère Enfant, Bron
  - Maladie Neuromusculaire de l'enfant - Service Maladies infectieuses et neurologie infantile - Hôpital Roger Salengro, Lille
  - Centre de référence Maladies Neuromusculaires Nantes-Angers - Hôtel Dieu, Nantes
  - I-Motion Institute - Trousseau Hospital, Paris
  - Neuropédiatrie - Service de Pédiatrie 1 - CHU Hautepierre, Strasbourg
  - Unité de neurologie pédiatrique - Hôpital des enfants, Toulouse
- Universitätsklinikum Essen (AöR) - Klinik für Kinderheilkunde I - Sozialpädiatrisches Zentrum, Essen, Germany

REFERENCES:
- [Derived] Chabanon A, Seferian AM, Daron A, Pereon Y, Cances C, Vuillerot C, De Waele L, Cuisset JM, Laugel V, Schara U, Gidaro T, Gilabert S, Hogrel JY, Baudin PY, Carlier P, Fournier E, Lowes LP, Hellbach N, Seabrook T, Toledano E, Annoussamy M, Servais L; NatHis-SMA study group. Prospective and longitudinal natural history study of patients with Type 2 and 3 spinal muscular atrophy: Baseline data NatHis-SMA study. PLoS One. 2018 Jul 26;13(7):e0201004. doi: 10.1371/journal.pone.0201004. eCollection 2018. PMID 30048507